CLINICAL TRIAL: NCT00776178
Title: Feasibility Study: Follow-Up of Bladder Cancer Patients From the New England Study of Environment and Health
Brief Title: Follow-Up of Bladder Cancer Patients From the New England Study of Environment and Health
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909007; 09-C-N007
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer
Keywords: Survival Study; Bladder Cancer; Cancer Recurrence; Tumor Markers/Heterogeneity
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Background:

* Bladder cancer often recurs after treatment and patient survival varies greatly.
* More knowledge is needed about factors that can help identify patients who are at greater risk of disease recurrence and progression to minimize the need for screening and to help guide treatment.
* The New England Study of Environment and Health (NESEH), conducted by the departments of health in Maine, New Hampshire and Vermont, the Dartmouth Medical School and the NIH, examined the relationship between health and environmental factors such as smoking, diet and water quality in New England. This study provides an opportunity to learn more about patients with bladder cancer.
* Before launching a full-scale follow-up study on bladder cancer, it is necessary to determine the feasibility of obtaining needed follow-up information from patients enrolled in the NESEH.

Objectives:

-To determine the completeness and quality of information about treatment, recurrence, and progression that can be obtained for patients from their medical records.

Eligibility:

-Participants from the NESEH study who are residents of Maine and who were diagnosed with bladder cancer between 2001 and 2003.

Design:

* Determine the vital status of NESEH bladder cancer patients.
* Select a sample of 40 living and 18 deceased patients.
* Interview patients or their next of kin by telephone for about 30 to 45 minutes to update exposure information, obtain names and addresses of all hospitals and physicians they have seen since diagnosis, and obtain authorization to access medical records.
* Obtain and abstract medical records.

DETAILED DESCRIPTION:
Background:

* Bladder cancer is a highly recurrent disease with substantial variability in survival.
* Patients currently undergo repeated cystoscopy for many years after diagnosis.
* There is a need to identify prognostic markers of recurrence and progression to minimize the need for routine screening and to identify patients who should be treated more aggressively.
* The New England Study of Environment and Health (NESEH), a population-based case control study of 1,213 patients in Maine (ME), Vermont (VT), and New Hampshire (NH), provides an excellent opportunity study the clinical, host-genetic, and environmental determinants of prognosis.
* Before launching a full-scale follow-up study, we need to determine the feasibility of following a population-based case series and of obtaining patient-related (vital status, exposures) and tumor-related (recurrence, progression, pathology) information.

Objectives:

To determine:

* The completeness and quality of information that can be obtained for each patient. The most important issue is the extent to which medical records from private physicians will be needed, and whether private physicians are cooperative.
* Our ability to identify next-of-kin (NOK) of deceased patients.
* The proportion of patients (and NOK) that we can contact and enroll.
* The ability of NOK to provide information on exposures.

Eligibility:

-Bladder cancer patients from ME who participated in the original case-control study (ages 30-79, newly diagnosed with histologically-confirmed carcinoma of the bladder, including carcinoma in situ), excluding those diagnosed after 2003 (5 years of follow-up are needed).

Design:

* Conduct interviews with 40 living patients and the NOK of 9 deceased patients to update exposure information and find out where the patient received health care, the types of treatment received, and whether and when the disease recurred or progressed.
* For living patients or NOK that we are unable to locate (an estimated 10 living patients and 9 NOK), request medical records from health care providers (to see if physicians will provide records in the absence of an authorization form).
* Evaluate participant and physician response rates and the completeness of the medical history information obtained.
* We will proceed with the full study if we obtain sufficient medical information for 70% of the living patients.
* We will examine whether there were important issues related to deceased patients (e.g., NOK identification/enrollment, exposure assessment, access to medical records). If so, consider a simpler approach for this segment of the population (e.g., survival study based on NDI Plus and information available from the NESEH).

ELIGIBILITY:
* INCLUSION CRITERIA:

With the exceptions noted below, all bladder cancer patients who participated in the NESEH and were residents of ME when first diagnosed with bladder cancer will be eligible for this feasibility study. Patients were eligible for the NESEH if they met the following criteria:

* 30-79 years old at initial diagnosis
* Newly diagnosed with histologically-confirmed carcinoma of the urinary bladder (including carcinoma in situ) between September 1, 2001 and October 31, 2004

EXCLUSION CRITERIA:

We will exclude from the feasibility study the following NESEH case participants:

* 44 bladder cancer patients (7 percent) first diagnosed at one of seven hospitals located in remote areas of ME (Aroostook Medical Center, Calais Regional Hospital, Cary Medical Center, Down East Community Hospital, Houlton Regional Hospital, Northern Maine Medical Center, and Mount Desert Hospital); this is for cost considerations;
* Patients diagnosed fewer than 5 years before the feasibility study begins (i.e., after 2003)

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The New England Study of Environment and Health (NESEH), a population-based case control study of 1,213 patients in Maine (ME), Vermont (VT), and New Hampshire (NH), provides an excellent opportunity study the clinical, host-genetic, and environmental determinants of prognosis. Bladder cancer patients from ME who participated in the original case-control study (ages 30-79, newly diagnosed with histologically-confirmed carcinoma of the bladder, including carcinoma in situ), excluding those diagnosed after 2003 (5 years of follow-up are needed).
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2008-10-17; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
There is no intervention. We are looking at survival. | September 30, 2015
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Stella Koutros, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Herr HW. Natural history of superficial bladder tumors: 10- to 20-year follow-up of treated patients. World J Urol. 1997;15(2):84-8. doi: 10.1007/BF02201977. PMID 9144896
- [Background] Holmang S, Hedelin H, Anderstrom C, Johansson SL. The relationship among multiple recurrences, progression and prognosis of patients with stages Ta and T1 transitional cell cancer of the bladder followed for at least 20 years. J Urol. 1995 Jun;153(6):1823-6; discussion 1826-7. PMID 7752327
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208